CLINICAL TRIAL: NCT02092519
Title: A Prospective Multi-center Randomized Study of the Difference in Diagnostic Yield Between EUSFNA Needles With and Without a Side Port in Pancreatic Masses
Brief Title: RCT: Difference in Diagnostic Yield Between EUSFNA Needles With and Without a Side Port in Pancreatic Masses
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Changi General Hospital (Other)
Collaborators: Asan Medical Center (Other); National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: ATL2012/312/E
Record Dates: First submitted 2014-02-20; First posted 2014-03-20 (Estimated); Last update posted 2015-07-29 (Estimated); Status verified 2015-07

CONDITIONS: Pancreatic Neoplasm; Pancreatic Diseases
Keywords: EUSFNA; endoscopic ultrasound; pancreatic masses
MeSH Terms: conditions — Pancreatic Neoplasms; Pancreatic Diseases | interventions — Needles

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Needle without sideport (NA-220H-8022) (Active Comparator): EUSFNA using needle without sideport (NA-220H-8022)
  Interventions: Device: Needle with sideport (NA-230H-8020)
- Needle with sideport (NA-230H-8020) (Active Comparator): EUSFNA using needle with sideport (NA-230H-8020)
  Interventions: Device: Needle without sideport (NA-220H-8022)

INTERVENTIONS:
Device: Needle with sideport (NA-230H-8020) — EUSFNA using needle with sideport
  Arms: Needle without sideport (NA-220H-8022)
Device: Needle without sideport (NA-220H-8022) — EUSFNA using needle without sideport
  Arms: Needle with sideport (NA-230H-8020)

SUMMARY:
Background: EUS-guided fine needle aspiration (EUSFNA) is a well established technique for tissue acquisition and diagnosis with excellent safety profile. The overall diagnostic yield of EUSFNA exceeds 80%, with higher rates in EUSFNA of lymph nodes, where rates of >90% may be expected, as compared to pancreatic masses, where lower diagnostic rates were reported. To maximize the diagnostic yield, at least 3 needle passes are required for lymph nodes and at least 4 passes for pancreatic masses. Olympus has recently made commercially available a new 22 gauge FNA needle (EZ Shot 2 with side port) with a side port at the needle tip. The theoretical basis for introduction of the side port is to increase the diagnostic yield. Preliminary unpublished retrospective data suggested the yield might be raised. However, there are no prospective multicenter randomized controlled studies to ascertain the validity of the assumption.

Aim: To determine whether there is a difference in diagnostic yield between EZ-Shot 2 and EZ-Shot 2 with side port in patients with pancreatic masses for evaluation.

Methods: Patients with pancreatic masses referred for EUSFNA will be recruited prospectively and randomized to either EZ-Shot 2 or EZ Shot 2 with sideport for the first puncture, and then the alternative needle will be used for repeated punctured. The cytological and diagnostic yield at first pass for both needles will be compared.

Clinical significance: This will determine whether the new needle design can further improve the diagnostic yield of EUSFNA of pancreatic masses.

DETAILED DESCRIPTION:
Background Endoscopic ultrasound (EUS) and EUS-guided fine needle aspiration (EUSFNA) are well established techniques in clinical practice. In routine gastrointestinal endoscopy such as gastroscopy, only the mucosal layer of the digestive tract is visualized. In the case of EUS, an ultrasonic transducer located at the tip of the echoendoscope allows the endoscopist to visualize the wall of gastrointestinal tract as a series of definable layers corresponding to histology, rather than as a single entity, and also enables detailed images of areas outside of the digestive tract, such as intra-abdominal lymph nodes, and solid organs such as liver, pancreas to be seen. EUS has a significant clinical impact because it allows assessment of submucosal GI lesions, loco-regional staging of gastrointestinal malignancy, tissue diagnosis by EUSFNA and staging of pancreaticobiliary lesions, non-small-cell lung carcinoma, and mediastinal disease. EUSFNA is a minimally invasive technique of tissue acquisition under EUS guidance. A FNA needle is inserted through the accessory channel of a curvilinear echoendoscope. Both the target lesion and the needle tip are visualized under real time ultrasound guidance, and any potential intervening vessels can be excluded by turning on the Doppler mode prior to needle puncture. The lesion is then punctured under real-time ultrasonic guidance and material aspirated by the needle for cytological assessment.

In prospective trials, EUSFNA has been clearly established to be an important diagnostic tool, with excellent safety profile. The overall diagnostic yield of EUSFNA should exceed 80%, with higher rates in EUSFNA of lymph nodes, where rates of >90% may be expected, as compared to pancreatic masses, where lower diagnostic rates were reported. The somewhat lower rates for solid pancreatic lesions compared to lymph nodes could be due to the underlying desmoplastic changes associated with pancreatic malignancies.

EUSFNA may be performed with rapid on site cytopathological assessment (ROSE) of the aspirated material to guide the number of needle passes being performed. In most practices, rapid on site cytopathological assessment is not feasible and it has been recommended that in such situation, in order to maximize the diagnostic yield, at least 3 needle passes should be performed for lymph nodes and at least 4 passes should be performed for pancreatic masses. Even without onsite cytopathological assessment, excellent results with greater than 90% diagnostic yield have been reported by expert centers.

Needles for EUSFNA are available from four manufacturers, namely Cook Endoscopy, Boston Scientific, Olympus Corporation and Mediglobe. The available needle diameters are 25, 22 and 19 gauge. These needles have a sharp tip for puncturing and a hollow core for aspiration after the puncture. The hollow needle core is covered by a stylet which is withdrawn after the puncture to facilitate aspiration. Aspiration is usually facilitated by application of suction using a syringe which is attached to the entry port of the hollow core of the needle, after the stylet has been withdrawn, although it must also be acknowledged that there are endoscopists who prefer to apply no suction in order to reduce the possibility of bloody aspirates. Olympus has recently made commercially available a new 22 gauge FNA needle with a side port at the needle tip. The theoretical basis for introduction of the side port is to facilitate the process of fine needle aspiration, and to increase the diagnostic yield. There have been preliminary unpublished retrospective data that suggested the yield might be raised. However, there are no prospective multicenter randomized controlled studies to ascertain the validity of the assumption. Currently two needles with similar designs, apart from absence and presence of side port, are available from Olympus Corporation. These are the EZ-Shot 2 (model: NA-220H-8022) and EZ-Shot 2 with side port (NA-230H-8022)

Aim The aim of this prospective randomized study is to determine whether there is a difference in diagnostic yield between EZ-Shot 2 (model: NA-220H-8022) and EZ-Shot 2 with side port (NA-230H-8022) in patients with pancreatic masses for evaluation.

Materials and methods

1. Setting and trial design:

   Setting: International; multicenter. Trial design: Randomized prospective comparative study.
2. Subjects:

   Inclusion criteria: 1) all patients referred for EUSFNA of pancreatic masses; 2) informed consent is obtained for performance of EUSFNA.

   Exclusion criteria: 1) presence of active gastrointestinal bleeding; 2) presence of coagulopathy as defined by platelet count <50000/mm3 or/ and international normalized ratio >1.5; 3) the current use of thienopyridines (e. g. clopidogrel) in patents requiring anti-platelet therapy; 4) absence of procedural informed consent.
3. Informed Consent:

   The protocol will be approved by local Institutional Review Board. Patients will be giving informed consent for the procedure.
4. Interventions:

   Randomization: Randomization of the needle used for initial puncture will be carried in blocks of 5 with equal assignment to the EZ-Shot 2 (model: NA-220H-8022) and EZ-Shot 2 with side port (NA-230H-8022) needles. Once the first 2 punctures have been performed, the alternative needle will be used to obtain the subsequent needle passes.

   EUS and EUSFNA technique: EUS and EUS will be performed using a curvilinear echoendoscope according to standard techniques9 by a credentialed endoscopist or under the direct supervision of a credentialed endoscopist in the case of procedures performed by trainees. The patient will either undergo the procedure without sedation, under sedation or under general anesthesia as clinically indicated. As per standard technique, the lesion is visualized using EUS, and then the 22gauge EUSFNA needle (depending on randomization either NA-220H-8022 or NA-230H-8022) is introduced into the accessory channel of the echoendoscope and the lesion is punctured under real time ultrasonic guidance. After withdrawal of the stylet and application of suction by attachment of a syringe with negative pressure, the needle is moved to and fro within the lesion for approximately 30 seconds, and then the needle is withdrawn and the material aspirated is expressed onto glass slides by reinsertion of the stylet and direct smears are made either by the endoscopist or cytotechnician. This process is repeated once using the first needle. The alternative needle is then used to make 2 further punctures..

   Preparation of aspirated material and definition of cellular adequacy and diagnostic yield10,11: The material aspirated is expressed onto glass slides by reinsertion of the stylet and direct smears are made either by the endoscopist or cytotechnician. After expressing the cellular material onto glass slides, half the slides will be air-dried and half will be alcohol fixed (95% ethanol) for subsequent cytological assessment. When no further material can be expressed, the residual contents of the needle are flushed with 5 to 10 mL of sterile saline solution into a balanced salt solution. After flushing the needle, the outside of the needle and the stylet are vigorously wiped with saline solution-soaked sterile gauze to reduce cross contamination between passes.

   An adequate specimen is defined as the clear presence of target organ cells. In the case for the pancreas there must be at least 4 clusters of pancreatic acinar cells with or without the presence of malignant-appearing cells. A cytopathologist blinded to the needle used for FNA, will characterized each individual needle pass for assessment of adequate cellularity (0 [inadequate] or 1 [adequate]) and a diagnosis of malignancy (insufficient, normal, "suspicious," malignant). . The diagnosis arrived at for each needle pass will be compared with the final diagnosis which will be based on composite of cytology, histology and clinical course. The EUSFNA findings will be classified as 1) inadequate for diagnosis; 2) true positive for malignancy; 3) true negative for malignancy; 4) false positive for malignancy; 5) false negative for malignancy.
5. Statistics Sample size: As this is an exploratory study, a sequential trial design will be used to determine the ideal sample size. For the initial assessment, a total of 30 pancreatic masses will be targeted. Dependent on the outcome and trend, this may be further increased to 100 cases.

   Outcome variables:

   Primary 1. Compare 1st pass cellular adequacy rate each needle: 2. Compare the overall cellular adequacy rate each needle 3. Compare the overall diagnostic accuracy rate between both needles 4. Compare 1st pass diagnostic accuracy adequacy rate of each needle
6. Timetable of work Complete study within 6 months, but may extend to 24 months

ELIGIBILITY:
Inclusion criteria:

* all patients referred for EUSFNA of pancreatic masses
* informed consent is obtained for performance of EUSFNA.

Exclusion criteria:

* presence of active gastrointestinal bleeding
* presence of coagulopathy as defined by platelet count <50000/mm3 or/ and international normalized ratio >1.5
* the current use of thienopyridines (e. g. clopidogrel) in patents requiring antiplatelet therapy8
* absence of procedural informed consent.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-04; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
diagnostic accuracy | within 1 month after EUSFNA and cytological assessment
  Compare the overall diagnostic accuracy rate between both needles

CONTACTS AND LOCATIONS:
Overall Officials: Tiing Leong Ang, MD, Principal Investigator — Changi General Hospital
Locations (1):
- Changi General Hospital, Singapore, Singapore, Singapore

REFERENCES:
- [Background] Polkowski M, Larghi A, Weynand B, Boustiere C, Giovannini M, Pujol B, Dumonceau JM; European Society of Gastrointestinal Endoscopy (ESGE). Learning, techniques, and complications of endoscopic ultrasound (EUS)-guided sampling in gastroenterology: European Society of Gastrointestinal Endoscopy (ESGE) Technical Guideline. Endoscopy. 2012 Feb;44(2):190-206. doi: 10.1055/s-0031-1291543. Epub 2011 Dec 16. PMID 22180307
- [Background] Dumonceau JM, Polkowski M, Larghi A, Vilmann P, Giovannini M, Frossard JL, Heresbach D, Pujol B, Fernandez-Esparrach G, Vazquez-Sequeiros E, Gines A; European Society of Gastrointestinal Endoscopy. Indications, results, and clinical impact of endoscopic ultrasound (EUS)-guided sampling in gastroenterology: European Society of Gastrointestinal Endoscopy (ESGE) Clinical Guideline. Endoscopy. 2011 Oct;43(10):897-912. doi: 10.1055/s-0030-1256754. Epub 2011 Aug 12. PMID 21842456
- [Derived] Ang TL, Kwek AB, Seo DW, Paik WH, Cheng TY, Wang HP, Lau J. A prospective randomized study of the difference in diagnostic yield between endoscopic ultrasound-guided fine-needle aspiration (EUSFNA) needles with and without a side port in pancreatic masses. Endosc Int Open. 2015 Aug;3(4):E329-33. doi: 10.1055/s-0034-1391964. Epub 2015 May 26. PMID 26356802